CLINICAL TRIAL: NCT01995903
Title: Developing a Discrimination Model to Diagnose ALS Using Advanced MRI Techniques
Brief Title: Developing a Discrimination Model to Diagnose ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00061126
Record Dates: First submitted 2013-11-04; First posted 2013-11-27 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amyotrophic lateral sclerosis (Experimental): Clinical examination for ALS(amyotrophic lateral sclerosis) and subjects with lower motor neuron signs will be completed. These subjects will undergo MRI (magnetic resonance imaging) scans of the brain to assess neurological conditions.
  Interventions: Diagnostic Test: MRI(magnetic resonance imaging)
- Healthy controls (MRI) (Active Comparator): These subjects will undergo MRI (magnetic resonance imaging) scans of the brain to compare against diseased subjects.
  Interventions: Diagnostic Test: MRI(magnetic resonance imaging)

INTERVENTIONS:
Diagnostic Test: MRI(magnetic resonance imaging) — Subjects with amyotrophic lateral sclerosis and lower neuron motor skills and healthy subjects will undergo an MRI(magnetic resonance imaging)scans of the brain to assess neurologic condition. The brain scans will take approximately 60 minutes to complete.

SUMMARY:
To combine several brain imaging techniques to develop a new diagnostic test to help with earlier diagnosis of amyotrophic lateral sclerosis.

DETAILED DESCRIPTION:
Early diagnosis and lack of understanding of the pathophysiology of ALS remain a significant obstacle to making a timely intervention to help patients suffering from this fatal disease. We envision a future in which neuroimaging techniques will be a critical tool in the diagnostic work-up of ALS. Advanced neuroimaging techniques offer great potential in identifying central nervous system metabolite and cellular alterations in ALS. We propose an innovative approach to combine complementary advanced MRI techniques to interrogate brain chemistry (MRS), brain microstructure (DTI) and brain function (fcMRI) and develop a clinically relevant discriminatory disease model.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. subjects with ALS (amyotrophic lateral sclerosis)
3. healthy subjects -

Exclusion Criteria:

1. Active substance abuse
2. Has co-morbid psychiatric disease
3. Has opportunistic CNS (central nervous system) infection
4. Has a history of head injury
5. Has a contraindication for MRI (e.g. cardiac pacemaker, ferromagnetic or metallic implants)
6. Pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Developing a Discrimination Model to Diagnose ALS | 5 years
  We will measure brain fractional anisotropy (unitless) using diffusion tensor imaging of ALS patients and compare these to corresponding measures in healthy control subjects as well as patients with lower motor neuron signs only.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Foerster, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No